CLINICAL TRIAL: NCT05739357
Title: Perioperative Complications and Cognitive Outcome in Carotid Thrombendarterectomy With Multimodal Monitoring Cerebral Perfusion Optimisation
Brief Title: Neurocognitive Function After Carotid Thrombendarterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Tina Tomic Mahecic, Consultant anesthesiologist, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UHCZagreb 02/21 AG
Record Dates: First submitted 2022-12-30; First posted 2023-02-22 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Carotid Stenosis; Postoperative Cognitive Dysfunction; Neurological Impairment
Keywords: CEA ACI; cognitive tests; BHI; NIRS; TCD; EEG
MeSH Terms: conditions — Carotid Stenosis; Postoperative Cognitive Complications; Neurologic Manifestations | interventions — Spectroscopy, Near-Infrared; Electroencephalography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cerebral perfusion monitoring (Active Comparator): Multimodal monitoring includes cerebral oxygenation (with NIRS) and EEG (with SEDLINE). During the carotic clamp, if cerebral oxygenation decreased for more than 12 % on the operating side from the baseline value, simple interventions as, increasing arterial blood pressure, increasing arterial carbon dioxide tension or increasing oxygen inspiration concentration will be performed.
  Interventions: Device: NIRS, EEG
- Control (No Intervention): The control arm does not have any monitor of cerebral perfusion and oxygenation, during the carotic clamp only intervention is regulating arterial blood pressure values.

INTERVENTIONS:
Device: NIRS, EEG — During the carotic clamp, if cerebral oxygenation decreased for more than 12 % on the operating side from the baseline value, simple interventions as, increasing arterial blood pressure, increasing arterial carbon dioxide tension or increasing oxygen inspiration concentration will be performed.
  Other Names: cerebral oximetry
  Arms: Cerebral perfusion monitoring

SUMMARY:
Previous studies did not reach a consensus on the influence of the type of anesthesiologic procedure and monitoring, during carotid thrombendarterectomy, on perioperative complications and cognitive outcomes. The aim of this study is the optimization of brain perfusion during the vascular carotid clamp using multimodal monitoring. We assume that standardized monitoring techniques and a better selection of cognitive tests will allow a more accurate assessment of subclinical cognitive deficits.

DETAILED DESCRIPTION:
ABSTRACT:

AIM OF THE STUDY: Effect of perioperative multimodal monitoring with transcranial doppler (TCD), near-infrared spectroscopy (NIRS), and Electroencephalography (EEG) in patients for carotid thrombendarterectomy (CEA) on perioperative complications and cognitive functions.

PATIENTS AND METHODS: The prospective study will analyze 80 consecutive patients with an asymptomatic and symptomatic (transitory ischemic attack, TIA, in anamnesis) stenosis of the internal carotid artery in which CEA is indicated in general anesthesia. Cognitive tests will be analyzed for all patients preoperatively, first and eighth day postoperatively, and after 8 weeks. Breath-holding index (BHI) will be measured preoperatively and postoperatively. The first group of patients (n = 40) will have expanded intraoperative monitoring involving TCD, NIRS, and EEG, and the control group (n = 40) will have only standard anesthetic monitoring.

EXPECTED CONTRIBUTION OF THE STUDY: Previous studies did not agree on the influence of the type of anesthesiologic procedure and monitoring of perioperative complications and cognitive outcomes. We assume that standardized monitoring techniques and a better selection of cognitive tests will allow a more accurate assessment of the effect.

ELIGIBILITY:
Inclusion Criteria:

* patients with The North American Symptomatic Carotid Endarterectomy Trial (NASCET) stenosis of more than 70%
* symptomatic stenosis
* asymptomatic stenosis
* elective surgery patients
* signed informed consent
* initial MoCa test equal and more than 22

Exclusion Criteria:

* who refuse to participate
* previous stroke in anamnesis
* patient without bone window for BHI measurements
* comorbidities with aphasia and plegia, and the impossibility to solve cognitive tests

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Change in measurements (result is in numbers) done at four time points (before surgery, day after the surgery, on 7th day and after 8 weeks
  A widely used screening assessment for detecting cognitive impairment. It was validated in the setting of mild cognitive impairment, and has subsequently been adopted in numerous other settings clinically. This test consists of 30 points and takes part in 10 minutes from the individual. The Montreal test is performed in seven steps. The basics of this test include short-term memory, executable performance, attention, focus and more.
Trail making test (TMT) 1 | Changes in measurements (results are in seconds) done at four time points (before surgery, day after the surgery, on 7th day and after 8 weeks
  Neuropsychological test that involves visual scanning and working memory. In the TMT-1 (rote memory) the subject is instructed to connect a set of 25 dots as quickly as possible (time is measured in seconds).
Trail making test (TMT) 2 | Changes in measurements done at four time points (before surgery, day after the surgery, on 7th day and after 8 weeks
  TMT-2 (executive functioning) is a neuropsychological test that involves visual scanning and working memory. In this test the dots go from 1 to 13 and include letters from A to L.
Month backwards test (MBT) | changes in measurements done at four time points (before surgery, day after the surgery, on 7th day and after 8 weeks
  It is a rapid (< 2 min) and simple to administer test of cognitive function that is widely used at the bedside. The test requests the subject to recite the months of the year in reverse order starting with December, until the subject reaches January.

SECONDARY OUTCOMES:
Difference in brain reactivity measured by Breath holding index | 8 weeks
  Difference in breath holding index before surgery , after the surgery and after eight weeks as a surrogate of brain perfusion in both groups of patients

CONTACTS AND LOCATIONS:
Overall Officials: Tina Tomic Mahecic, Principal Investigator — UHC Zagreb
Locations (1):
- UHCZagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No